CLINICAL TRIAL: NCT03598725
Title: Beijing Children's Hospital, Capital Medical University
Brief Title: Low-dose ITI Strategy for Children in Hemophilia A With High-titer Inhibitor and Poor ITI Risk in China
Acronym: HA-LD-ITI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Runhui WU, Capital Medical Univercity, Beijing Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-ITI-20180123
Record Dates: First submitted 2018-01-23; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hemophilia A With Inhibitor
MeSH Terms: interventions — Factor VIII; Prednisone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ITI strategy (Experimental): The low-dose ITI was Coagulation Factor VIII (50IU/kg, every other day) alone or combined with prednisone (2mg Kg-1/day, one month, then taper in three months) depending on the tendency of inhibitor, and Rituximab (375mg/square meter every week for 4 weeks) when the inhibitor titer ≥40BU/ml before or during ITI.Inhibitor and hemorrhage should be retested and recorded periodically.
  Interventions: Drug: Coagulation Factor VIII; Drug: Prednisone; Drug: Rituximab

INTERVENTIONS:
Drug: Coagulation Factor VIII — Domastic plasma derived factor FVIII (with intermidiate vWF) 50IU/kg every other day
Drug: Prednisone — 2mg/kg every day for 4 weeks then typering in 3 months
Drug: Rituximab — 375mg/Square meter for consecutive 4 months

SUMMARY:
The study start on January 18, 2017. The Severe(FⅧ<1%) and moderate hemophilia A (FⅧ1%～5%)children with high titer inhibitor(historical peak inhibitor titer≥5BU ) combining with poor ITI risk(s) were enrolled. The low-dose ITI was alone or combined with immunosuppression.

DETAILED DESCRIPTION:
Poor risk(s) includes:①peak historical inhibitor titer≥200BU ②inhibitor titer≥10BU before ITI initiation ③peak inhibitor titer during ITI≥200BU ④time to titer decline to<10BU before ITI≥24 months ⑤age≥8 years at start of ITI ⑥ITI initiated ≥5 years after inhibitor diagnosis ⑦interruptions in ITI≥2 weeks in duration. The low-dose ITI strategy consist of FⅧ（25-50IU/kg）alone or combining with immunosuppression: prednisone and Rituximab when the inhibitor titer ≥40BU ml/ml before or during ITI.

ELIGIBILITY:
Inclusion Criteria:

* Males
* from 1 to 14 years old
* severe or moderate hemophilia A;
* inhibitors positive before ITI started.

Exclusion Criteria:

* Females
* <1 or >14 years old
* hemophilia B or mild haemophilia A;
* inhibitor negative before ITI started.

Ages: 1 Year to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 2 years
  Success rate

SECONDARY OUTCOMES:
Annualized Bleeding Rate | 2 year
  How many times for all types of bleeding
Annualized Joint Bleeding Rate | 2 year
  How many times for joint bleeding
Success time | 2 years
  How long to success

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Z, Tang Y, Chen Z, Liu G, Yao W, Li G, Cheng X, Peng Y, Cai S, Cui C, Ai D, Zhang J, Poon MC, Zhang W, Wu R. Outcomes of immune tolerance induction with rituximab to eradicate high-titer inhibitor of hemophilia A: depicted by exponential decay model and the gene expression profile of different outcomes by RNA-sequencing. J Thromb Haemost. 2025 Aug;23(8):2436-2448. doi: 10.1016/j.jtha.2025.04.015. Epub 2025 Apr 24. PMID 40286913